CLINICAL TRIAL: NCT02957734
Title: The Use of LAVA Ultimate Restorations in a Full Occlusal Rehabilitation for Patients With Severe Tooth Wear
Brief Title: Full Occlusal Rehabilitation for Patients With Severe Tooth Wear Using Indirect Composite Restorations
Acronym: NTWP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: 3M ESPE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTWP-LAVA2016
Record Dates: First submitted 2016-10-12; First posted 2016-11-08 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Tooth Wear; Dental Restoration Failure; Dental Restoration Wear
Keywords: Vertical dimension of occlusion; Direct composite restorations; Indirect composite restorations; Tooth wear; Failure; Quality of Life
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LAVA Ultimate restorations (Experimental): For rehabilitation of the severely worn teeth, teeth are prepared (based on Minimal Invasive procedures), scanned using an intra-oral 3D-scanner (TrueDef, 3M), a digital wax-up model is made and finally restorations are milled from a pre polymerized block of resin (LAVA Ultimate). These indirect restorations are then adhesively cemented on the teeth (Relyx Ultimate, 3M). Teeth on which no indirect restoration could be made/designed a direct composite restoration was made using Filtek Supreme XTE in combination with Scotchbond Universal. Furthermore, all anterior veneer restorations are made of direct composite restorations (Filtek Supreme XTE in combination with Scotchbond Universal).
  Interventions: Procedure: Rehabilitation of severely worn dentitions

INTERVENTIONS:
Procedure: Rehabilitation of severely worn dentitions — Patients with severely worn dentition and functional problems are included in this study. Teeth are rehabilitated using indirect composite resin restorations in an increased vertical dimension of occlusion in order to optimize function and esthetics.

SUMMARY:
LAVA Ultimate composite restorations will be used as restorative material to reconstruct severely worn dentitions.

DETAILED DESCRIPTION:
Standard dental treatment will be provided to the patients with severely worn dentitions. Treatment is based on the principles of 'minimally invasive treatment techniques'.

Main difference with the 'standard' treatment protocol and the standard procedure of placing composite restorations is the fully digital workflow. In the traditional workflow a silicon impression is made, after which the dental technician produces the (indirect) composite restorations in by hand. These restorations are then adhesively cemented on the teeth by the dentist. In the fully digital workflow, digital 3D-scans are made using the 3D LAVA scanner (3M ESPE). Based on these digital 3D-images a digital wax-up is made by the dental technician after which all composite restorations (uplays and backings) are designed digitally before being milled and finally adhesively cemented on the teeth by the dentists. An important benefit for the patients is the rehabilitation of their worn dentitions. Functionality (teeth are less sensitive, improved chewing ability, a better occlusal stability, etc) and aesthetics will be improved immediately after finishing the treatment. Moreover, the estimated treatment time will be less (estimated treatment time approx. 12hours) than the traditional methods when using the standard treatment protocol (estimated treatment time approx. 18hours).

Another potential benefit is a better control and more predictable results by using 3D-images with the pre-designed computer simulation.

A risk of these indirect composite resin restorations is the unknown survival rate compared to other indirect as well as to direct application technique

ELIGIBILITY:
Inclusion Criteria:

* Generalized severe tooth wear
* Presence of functional problems
* Necessary increase of vertical dimension of occlusion (VDO) of ≥3 mm at location of first molars
* No edentulous space in need for treatment in the anterior region in upper and lower jaw
* A minimum of three posterior teeth (premolars and molars) per quadrant

Exclusion Criteria:

* ASA 4
* Functional problems (mouth opening < 5cm, severe Tempero Mandibular Dysfunction)
* Severe periodontitis (DPSI = 4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Surival of indirect composite restorations in patients treated for severe tooth wear | Failures one year after placement
  Percentage of failed restorations and the clinical success of the restorations and the relation of the failures with etiological factors

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Opdam N, Skupien JA, Kreulen CM, Roeters J, Loomans B, Huysmans MD. Case Report: A Predictable Technique to Establish Occlusal Contact in Extensive Direct Composite Resin Restorations: The DSO-Technique. Oper Dent. 2016 Sep;41(S7):S96-S108. doi: 10.2341/13-112-T. Epub 2016 Feb 26. PMID 26918925
- [Derived] Maier E, Crins L, Pereira-Cenci T, Bronkhorst E, Opdam N, Galler K, Loomans B. 5.5-year-survival of CAD/CAM resin-based composite restorations in severe tooth wear patients. Dent Mater. 2024 May;40(5):767-776. doi: 10.1016/j.dental.2024.03.001. Epub 2024 Mar 7. PMID 38458918